CLINICAL TRIAL: NCT00887653
Title: Changes in Lipid Profiles and Safety of Raltegravir Based Antiretroviral Therapy in HIV-1-infected Patients With Hyperlipidemia While on Current Standard Therapy
Brief Title: Changes in Lipids and Safety of Raltegravir in HIV+ Patients With Hyperlipidemia While on Current Standard Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Tufts Medical Center (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Aadia Rana, Assistant Professor of Medicine, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-09
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: HIV; Hyperlipidemia; Hypertriglyceridemia; HIV Infections
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia; HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental): This is a single arm study where HIV-infected individuals virologically suppressed on current regimen will be switched to raltegravir +optimized back ground regimen for 6 months
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — This will be a single arm study where subjects will be given the option to switch from their current regimen to raltegravir at 400mg twice daily.
  Other Names: Isentress

SUMMARY:
The success of combination antiretroviral therapy heralded a revolution in the treatment of HIV in the mid-1990s. However, severe treatment-associated side effects have been observed including diabetes and increased cholesterol which are linked to premature heart attacks. This effect has been described among many regimens containing protease inhibitors (PIs), as well as non-nucleoside reverse transcriptase inhibitors (NNRTIs). Raltegravir is a new medicine which has been shown to be potent and efficacious in suppression of the HIV. This study hopes to determine if switching from a PI or NNRTI to raltegravir will decrease cholesterol in subjects with high cholesterol and well controlled HIV. In addition, the study aims to confirm that raltegravir is safe and well tolerated. It also seeks to confirm if raltegravir will have similar anti-HIV activity compared with the patient's previous regimen.

The study will last 6 months and will involve 20 subjects. HIV-1 infected men and women on PIs or NNRTIs for at least 12 months before study entry with well controlled HIV will be recruited.

Hypotheses:

1. Patients with elevated lipid levels while on combination antiretroviral therapy with PIs or NNRTIs will experience an improvement in lipid levels after switching their PI or NNRTI to a raltegravir based regimen.
2. Raltegravir will be safe and well tolerated.
3. Raltegravir will have similar antiretroviral activity compared with the prior regimen.

Primary Objective:

To demonstrate an improvement in lipid profile (triglycerides or LDL) in subjects switched to raltegravir from PIs or NNRTIs at 2, 3, and 6 months after study entry.

Study Design: Subjects will be given the option to switch from their current regimen to raltegravir at 400mg twice daily. Those who consent, will receive raltegravir provided by the study for 6 months. At entry, the subjects will undergo a complete physical exam and thereafter targeted exams at each visit. Labs will be drawn as part of clinical care at 2, 3, and 6 months. Some of the blood will be stored for later analysis. Also, the subjects will answer regular surveys on drug toxicity and quality of life. Their cholesterol level will be compared before and after the study. At the end of the study, the participants may choose to continue on raltegravir if they desire.

DETAILED DESCRIPTION:
The success of combination antiretroviral therapy heralded a revolution in the management of patients with HIV in the mid-1990s. Increasingly, severe treatment-associated metabolic side effects have been observed and linked to premature coronary artery disease. This effect has been described among many regimens containing protease inhibitors (PIs) as well as non-nucleoside reverse transcriptase inhibitors (NNRTIs).

Raltegravir is a novel HIV-1 integrase inhibitor which in a comparison study with efavirenz has been shown to be potent and efficacious in suppression of the HIV-1. Minimal side effects were reported which mainly included nausea, headache, dizziness, diarrhea, and insomnia.

Hypotheses:

1. Patients with elevated lipid levels while on combination antiretroviral therapy with PIs or NNRTIs will experience an improvement in lipid levels after switching their PI or NNRTI to a raltegravir based regimen.
2. Raltegravir will be safe and well tolerated.
3. Raltegravir will have similar antiretroviral activity compared with the prior regimen.

Primary Objective:

To demonstrate an improvement in triglycerides or LDL in subjects switched to raltegravir from PIs or NNRTIs at 2 months, 3 months, and 6 months after study entry.

Secondary Objectives:

To assess the immunologic and virologic outcomes in subjects switched to raltegravir from PIs or NNRTIs at 2, 3, and 6 months after entry.

Study Design:

This will be a single arm study where subjects will be given the option to switch from their current regimen to raltegravir at 400mg twice daily.

Primary endpoint: Change from baseline LDL and change from baseline triglycerides at 3 months, adjusted for BMI and smoking status.

The subjects' plasma viral load before and after switching will be compared with a paired t test at each time point.

The subjects' CD4+ T cell count will be compared with a paired t test before and after switching.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Fasting LDL>130 mg/dL
* Fasting triglycerides >250 mg/dL
* Plasma viral load below 50 copies/mL on current regimen for 6 months prior to study entry.
* No prior history of any NRTI resistance.

Exclusion Criteria:

* History of NRTI resistance mutations
* Need for medications that have drug interactions with raltegravir: dilantin, phenobarbitol and rifampin
* Unstable clinical condition, such as unstable cardiac disease, or cancer requiring ongoing chemotherapy or radiation therapy, or other medical condition which, in the opinion of the investigator, would preclude a subject from safely undergoing study procedures.
* Breast-feeding or pregnancy.
* Use of immunosuppressive medications within 60 days prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tashima, MD, Principal Investigator — The Miriam Hospital
Locations (2):
- United States (2):
  - Tufts University, Boston, Massachusetts
  - Miriam Hospital Immunology Clinic, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir Arm: This is a single arm study where HIV-infected individuals virologically suppressed on current regimen will be switched to raltegravir +optimized back ground regimen for 6 months
  raltegravir: This will be a single arm study where subjects will be given the option to switch from their current regimen to raltegravir at 400mg twice daily.
Period: Overall Study
Arm/Group | Raltegravir Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir Arm
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 52 [40 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Triglycerides
Description: Assess changes from baseline triglycerides at 3 months
Time Frame: 3 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Raltegravir Arm
Number analyzed (Participants) | 20
units on a scale | 125 [93 to 224]

2. Secondary Outcome: Proportion of Patients With Plasma Viral Load Below the Limit of Detection
Description: Assess proportion of patients with PVL below limit of detection at end of study.
Time Frame: 6 months
Population: One subject was prematurely discontinued from the study at week 12 due to detectable HIV-1 RNA of 57 copies/mL that was sustained at 61 copies on repeated measurement two weeks later.
Measure: Number; unit: proportion of participants
Arm/Group | Raltegravir Arm
Number analyzed (Participants) | 20
proportion of participants | 0

3. Primary Outcome: Change From Baseline Triglycerides
Description: Assess changes from baseline triglycerides at 6 months
Time Frame: 6 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Raltegravir Arm
Number analyzed (Participants) | 20
units on a scale | 120 [93.3 to 170.3]

ADVERSE EVENTS:
Arm/Group | Raltegravir Arm
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir Arm (N=20)
Virologic Failure (Immune system disorders) | 1 (1) — One subject was found at week 12 with HIV-1 RNA of 57 copies/mL; repeat with 61 copies. Genotype revealed no evidence of resistance. The subject was then initiated on darunavir/ritonavir regimen with subsequent re-suppression to <50 copies/mL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No